CLINICAL TRIAL: NCT05700279
Title: Preventing the Development of Chronic Pain: Treating PTSD at Acute Pain Onset
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 21092002
Record Dates: First submitted 2023-01-17; First posted 2023-01-26 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: PTSD; Chronic Pain
Keywords: PTSD; Chronic Pain; Acute Pain
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Chronic Pain; Acute Pain

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Stellate Ganglion Block Treatment (Active Comparator): Participants randomly assigned to the Stellate Ganglion Block (SGB) condition will receive 2 SGB treatments separated by 2 weeks.
  Interventions: Procedure: Stellate Ganglion Block
- Cognitive Processing Therapy (Active Comparator): Participants randomly assigned to the Cognitive Processing Therapy (CPT) condition will receive 1-week massed CPT treatment consisting of 10 CPT sessions given within a single 5-day period via telehealth.
  Interventions: Behavioral: Cognitive Processing Therapy
- Usual Care (No Intervention): Participants randomly assigned to the Usual Care condition will not receive any active intervention.

INTERVENTIONS:
Procedure: Stellate Ganglion Block — Stellate Ganglion Block (SGB) procedure involves an injection of a local anesthetic (0.5% ropivacaine) around the stellate ganglion (a bundle of nerves located at the base of the neck) to block the transmission of pain signals. The SGB injection is administered by an anesthesiologist.
  Arms: Stellate Ganglion Block Treatment
Behavioral: Cognitive Processing Therapy — Cognitive Processing Therapy (CPT) is a form of trauma-based talk therapy that will be conducted by clinical therapists. CPT can help people identify and challenge unhelpful trauma-related beliefs about themselves, others, and the world.
  Arms: Cognitive Processing Therapy

SUMMARY:
Although most people recover from acute pain (such as pain caused by injury, surgery, repetitive motion, or unknown causes), many people do not fully recover and will experience chronic pain. Untreated posttraumatic stress disorder (PTSD) appears to be a key risk factor for the transition from acute pain to chronic pain. However, few published studies have addressed the issue of preventing the transition from acute to chronic pain via PTSD reduction. This project will aim to test whether trauma-related PTSD symptoms can be reduced using either Stellate Ganglion Block (SGB) treatment or Cognitive Processing Therapy (CPT), and whether reducing PTSD symptoms can prevent the transition from non-injury based acute pain to chronic pain.

DETAILED DESCRIPTION:
Untreated PTSD appears to be a key risk factor for the transition from acute pain to chronic pain. Thus, reducing PTSD symptoms during an acute pain episode may potentially decrease the likelihood of transitioning to chronic pain. CPT is an evidence-based trauma-focused cognitive behavioral treatment that is hypothesized to reduce PTSD symptoms via reducing negative trauma-related cognitions about oneself, others, and the world. SGB treatment is an injection of a local anesthetic into the stellate ganglion, which is a bundle of nerves located at the base of the neck that is part of the sympathetic nervous system. Previous studies suggest that 1-week massed CPT and SGB treatment can both reduce the severity of PTSD symptoms in short periods of time via two distinct psychological and biological mechanisms.

This 4 year project will test study hypotheses in a sample of 345 individuals with PTSD symptoms who present to the presenting to the Rush University Medical Center ED or Rush's Primary Care and Preventive Medicine group with non-injury based acute pain. Participants will be randomly assigned to receive 1-week massed CPT, 2 SGB treatments, or usual care. All participants will complete identical self-report and/or clinician administered assessments at baseline (prior to randomization) and on study days 1, 7, 14, 21, 28, 56 (approximately 3 months after the initial ED presentation or Presentation to Preventive Medicine), and 112 (approximately 6 months after ED presentation or presentation to Preventive Medicine).

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 to 70 years
2. Ability to read and write English sufficiently to understand and complete study questionnaires and participate in interviews
3. Presenting to the Rush ED with acute pain without debilitating trauma
4. A primary acute pain site
5. Self-reported symptoms consistent with a diagnosis of PTSD
6. People with well-controlled diabetes or HIV/AIDS with chronic neuropathic pain will be included if their acute pain complaint at ED presentation is not due to neuropathic pain
7. Individuals with a history of psychotic or bipolar disorder that is currently well managed, have been treated for the condition for at least 3 months, are able to coherently answer interview questions, and are judged by study staff to be capable of participating in study
8. Current chronic illness that involves constant or frequent pain if their acute pain complaint at ED presentation is not due to the chronic illness. (case-by-case basis)
9. Current chronic pain from various sources if their acute pain complaint at ED presentation is not related to their current chronic pain. (case-by-case basis)

Exclusion Criteria:

1. Pain intensity great enough to impair concentration or capacity to understand instructions or the nature of being invited into a study as assessed by a member of the medical staff
2. Any injury or illness that precludes their ability to understand or follow instructions as assessed by a member of the medical staff
3. Self-reported history of chronic pain on presentation to the ED or documented in the electronic medical record (case-by-case basis)
4. Pain from traumatic event that is the source of their PTSD
5. Neurological disorder
6. Blood pressure greater than 160/100 mmHg
7. Taking anticoagulants or antiplatelet drugs other than aspirin
8. Pregnancy
9. Current alcohol or substance dependence
10. Anything that precludes interventions from being successful.
11. We will exclude people who are being treated for chronic or significant diseases such as rheumatoid disease, current influenza that may manifest temporary flu- related pain, and heart disease.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 345 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2027-02-01 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
Change in Patient-Reported Outcomes Measurement Information System (PROMIS) Pain Intensity | Through study completion, for an average of 6 months
  Intensity of chronic pain reported by subject. The PROMIS Pain Intensity scale consists of 3 questions with a 5-point response scale ranging from "Had no pain" -to "Very severe. " Participants are asked how intense their pain has been in the past 7 days. Higher scores indicate more intense pain.
Change in PTSD Checklist for Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (PCL-5) Self-Reported PTSD Symptoms | Through study completion, for an average of 6 months
  PCL-5 will be used to measure self-reported PTSD symptoms. The PCL-5 consists of 20 questions that ask how much a given symptom has bothered the participant within a specified time period. Each question has a 5 point response scale ranging from "not at all" (0) to "extremely" (4). Higher scores indicate greater PTSD symptom severity.

SECONDARY OUTCOMES:
Change in SCID-5 mood and anxiety disorder diagnoses | Through study completion, for an average of 6 months
  The Structured Clinical Interview for the DSM-5 (SCID-5) is a semi-structured interview measure for making DSM-5 diagnoses. The SCID-5 will be administered by a trained interviewer for assessment of mood and anxiety disorders.
Change in AUDIT-C Self-Reported Substance Use | Through study completion, for an average of 6 months
  The Alcohol Use Disorder Identification Test (AUDIT-C) is a self-report questionnaire consisting of 12 items that ask participants about the frequency of their alcohol and substance use both generally and within the past 2 weeks (14 calendar days).
Change in Patient-Reported Outcomes Measurement Information System (PROMIS) Pain Interference | Through study completion, for an average of 6 months
  Interference in daily activities attributed to chronic pain as reported by subjects. The PROMIS Pain Interference scale consists of 8 questions with a 5-point response scale ranging from "Not at all" to "Very much." Participants are asked how much in the past 7 days everyday activities were affected by their pain. Higher scores indicate more pain interference in daily activities.
Change in Patient-Reported Outcomes Measurement Information System (PROMIS) Depression (Short Form) | Through study completion, for an average of 6 months
  Degree of depressive symptoms reported by subject. The PROMIS Depression scale consists of 8 questions with a 5-point response scale ranging from "Never" to "Always." Participants are asked how often they felt depressive emotions in the past 7 days. Higher scores indicate more depressive emotions.
Change in Patient-Reported Outcomes Measurement Information System (PROMIS) Physical Function (Short Form) | Through study completion, for an average of 6 months
  Amount of physical activity reported by subject. The PROMIS Physical Function scale consists of 10 questions with a 5-point response scale ranging from "Without any difficulty" to "Unable to do." Participants are asked how much their pain affects their physical functioning. Higher scores indicate more inability to perform specific physical activities due to pain.
Change in Patient-Reported Outcomes Measurement Information System (PROMIS) sleep disturbance (short form) | Through study completion, for an average of 6 months
  Degree of sleep disturbance reported by subject. The PROMIS Sleep Disturbance scale consists of 8 questions with a 5-point response scale ranging from "Not at all" to "Very much." Participants are asked how much in the past 7 days their symptoms interfered with their sleep. Higher scores indicate more sleep disruptions.
Change in Patient-Reported Outcomes Measurement Information System (PROMIS) anxiety (short form) | Through study completion, for an average of 6 months
  Degree of anxiety symptoms reported by subject. The PROMIS Anxiety scale consists of 7 questions with a 5-point response scale ranging from "Never" to "Always." Participants are asked how often they experienced anxiety symptoms in the past 7 days. Higher scores indicate more anxiety symptoms.
Change in Patient-Reported Outcomes Measurement Information System (PROMIS) anger (short form) | Through study completion, for an average of 6 months
  Degree of anger reported by subject. The PROMIS Anger scale consists of 5 questions with a 5-point response scale ranging from "Never" to "Always." Participants are asked how often they experienced anger in the past 7 days. Higher scores indicate more frequent anger.
Change in Patient-Reported Outcomes Measurement Information System (PROMIS) Satisfaction with Social Roles | Through study completion, for an average of 6 months
  Satisfaction with social roles reported by subject. The PROMIS Satisfaction with Social Roles scale consists of 7 questions with a 5-point response scale ranging from "Not at all" to "Very Much." Participants are asked how satisfied they have felt with their performance in various social roles in the past 7 days. Higher scores indicate greater satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: John W Burns, PhD, Principal Investigator — Rush University Medical Center
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2024-06-03): https://cdn.clinicaltrials.gov/large-docs/79/NCT05700279/ICF_001.pdf